CLINICAL TRIAL: NCT04136626
Title: Digital Health Interventions for Obsessive Compulsive Disorder: A Randomized Controlled Trial
Brief Title: Digital Health Interventions for Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Koa Health B.V. (Industry)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Chief of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P001669
Record Dates: First submitted 2019-10-17; First posted 2019-10-23 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD; randomized controlled trial; digital health
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Perspectives OCD (Experimental): 12 week Smartphone-delivered cognitive behavioral therapy (CBT) for OCD.
  Interventions: Device: Perspectives OCD
- The Health and Well-Being Program (Active Comparator): 12 week health and well-being education
  Interventions: Device: The Health and Well-Being Program

INTERVENTIONS:
Device: Perspectives OCD — The app-delivered cognitive behavioral therapy (CBT) in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work) and behavioral skills (e.g., exposure and response prevention).
  Arms: Perspectives OCD
Device: The Health and Well-Being Program — The website includes 12 modules related to general health and well-being (e.g., sleep and nutrition). Each module contains educational information and questions about an indvidual's experience with the given topic.
  Arms: The Health and Well-Being Program

SUMMARY:
The investigators are testing two digital health interventions for obsessive compulsive disorder (OCD). The investigators hope that these digital health programs will increase access to treatment for OCD.

DETAILED DESCRIPTION:
The primary aims of this study are to test the feasibility, acceptability, and efficacy of two digital health interventions for adults with OCD recruited nationally. Eligible subjects (N=120) will be randomly assigned (50/50 chance) to 12 weeks of app-based CBT on their personal Smartphone or 12 weeks of web-based health and well-being education in addition to completing clinical assessments and questionnaires from home. All participants will have access to a coach to help guide them through their assigned program. Total participation time for the study is approximately 6 months, and all study appointments (5 total) occur over secure phone or video conference call.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Current diagnosis of primary obsessive compulsive disorder (OCD), based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), Mini International Neuropsychiatric Interview (MINI)
* Currently living in the United States

Exclusion Criteria:

* Psychotropic medication changes within 2 months prior to enrollment (Participants taking psychotropic medication must have been on a stable dose for at least 2 months prior to enrollment and not change medication during study period)
* Past participation in ≥4 sessions of cognitive behavioral therapy (CBT) for OCD
* Past use of a CBT for OCD app
* Current severe substance use disorder
* Lifetime bipolar disorder or psychosis
* Acute, active suicidal ideation as indicated by clinical judgment and/or a score ≥2 on the suicidal ideation subscale of the Columbia Suicide Severity Rating Scale (C-SSRS).
* Current severe comorbid major depression, as indicated by clinical judgment and/or a Quick Inventory of Depressive Symptomatology, self-report version (QIDS-SR), total score ≥ 21
* Current post-traumatic stress disorder (PTSD)
* Concurrent psychological treatment
* Does not own a supported mobile smartphone with a data plan
* Lack of technology literacy that would interfere with ability to engage with smartphone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wilhelm S, Greenberg JL, Jacoby RJ, Weingarden H, Hoeppner SS, Klare D, Snorrason I, Jaroszewski AC, McCoy TH, Harrison O. A randomized clinical trial of app cognitive behavior therapy vs. HealthWatch for obsessive compulsive disorder. NPJ Digit Med. 2025 Dec 15;8(1):800. doi: 10.1038/s41746-025-02230-9. PMID 41398456

RESULTS

PARTICIPANT FLOW:
Groups:
- Perspectives OCD: 12 week Smartphone-delivered CBT for OCD.
  Perspectives OCD: The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work) and behavioral skills (e.g., exposure and response prevention).
Period: Treatment Phase
Arm/Group | Perspectives OCD | The Health and Well-Being Program
Started | 60 | 60
Completed | 57 | 46
Not Completed | 3 | 14
Not completed — Withdrawal by Subject | 1 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 5
Period: 12-month Follow-up
Arm/Group | Perspectives OCD | The Health and Well-Being Program
Started | 57 | 46
3-month Follow-up | 52 | 41
Completed | 49 | 39
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perspectives OCD | The Health and Well-Being Program | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (14.7) | 41.1 (15.6) | 40.1 (15.1)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity, self-reported
  Participants
    Woman | 47 | 46 | 93
    Man | 10 | 11 | 21
    Transgender, non-binary, or questioning | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in the Health and Well-Being Program group did not provide data for sex at birth.
  Participants
    number analyzed (Participants) | 60 | 59 | 119
    Female | 50 | 48 | 98
    Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 57 | 52 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 48 | 44 | 92
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Education [Count of Participants; unit: Participants] — Population: One participant in the Health and Well-Being Program group did not provide data for education.
  Participants
    number analyzed (Participants) | 60 | 59 | 119
    High school graduate or less | 8 | 5 | 13
    Technical school / some college | 16 | 11 | 27
    College graduate | 21 | 15 | 36
    Graduate or professional school | 15 | 28 | 43
Marital status [Count of Participants; unit: Participants] — Population: One participant in the Health and Well-Being Program group did not provide data for marital status.
  Participants
    number analyzed (Participants) | 60 | 59 | 119
    Single, never married | 26 | 23 | 49
    Married | 23 | 28 | 51
    Partnered | 5 | 3 | 8
    Divorced / separated | 5 | 5 | 10
    Widowed | 1 | 0 | 1
Employment [Count of Participants; unit: Participants] — Population: One participant in each treatment group did not provide data for employment status.
  Participants
    number analyzed (Participants) | 59 | 59 | 118
    Employed full-time (>= 35 hours per week) | 27 | 35 | 62
    Employed part-time (< 35 hours per week) | 6 | 6 | 12
    Student | 6 | 6 | 12
    Unemployed | 11 | 5 | 16
    Retired | 5 | 2 | 7
    Homemaker | 4 | 5 | 9
Household income [Count of Participants; unit: Participants] — Population: Five participants did not provide income data (2 in Perspectives OCD, 3 in the Health and Well-Being Program group).
  Participants
    number analyzed (Participants) | 58 | 57 | 115
    $34,999 or less | 21 | 19 | 40
    $35,000 - 74,999 | 13 | 21 | 34
    $75,000 - 149,999 | 20 | 12 | 32
    $150,000 or more | 4 | 5 | 9
Duration of OCD [Mean (Standard Deviation); unit: years since onset] | 23.9 (15.3) | 26.5 (16.4) | 25.2 (15.8)
Current psychiatric comorbidities [Count of Participants; unit: Participants] — Clinician-assessed, based on the Miniature Neuropsychiatric Interview (MINI) Population: The diagnostic designation for generalized anxiety disorder was accidentally not assessed for one participant in the Health and Well-Being Program group.
  Participants
    Major depression | 9 | 8 | 17
    Panic disorder | 9 | 1 | 10
    Agoraphobia | 3 | 4 | 7
    Social anxiety disorder | 7 | 10 | 17
    Alcohol use disorder | 2 | 5 | 7
    Binge eating disorder | 1 | 2 | 3
    Generalized anxiety disorder: number analyzed (Participants) | 60 | 59 | 119
    Generalized anxiety disorder | 8 | 11 | 19
    Body dysmorphic disorder | 5 | 6 | 11
Number of comorbid axis I disorders [Count of Participants; unit: Participants] — We used the Mini International Neuropsychiatric Interview (M.I.N.I., English Version 7.0.2) to assess the most common psychiatric disorders and suicidality. The MINI was designed as a brief structured diagnostic interview to meet the need for a short but accurate structured psychiatric interview for clinical trials and studies. The MINI is a relatively short, structured clinical interview with very precise questions about psychological problems which require a yes or no answer from participants. In our study, the MINI was administered by trained clinicians.
  Participants
    None | 36 | 33 | 69
    1 | 12 | 11 | 23
    2 | 6 | 12 | 18
    3 or more | 6 | 4 | 10
Current psychotropic medication [Count of Participants; unit: Participants]
  None | 35 | 37 | 72
  Selective reuptake inhibitor (SRI) | 15 | 18 | 33
  Non-SRI antidepressant | 5 | 9 | 14
  Benzodiazepine | 6 | 1 | 7
  Antipsychotic | 1 | 0 | 1
  Other psychotropic medication | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Difference in OCD Symptom Severity at the End of Week 12
Description: Symptom severity for OCD was measured with the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), the gold-standard, semi-structured clinician-administered assessment of OCD severity. It contains 10 items ranging from 0 to 4, which are summed to generate a total score (range 0 to 40). Higher scores indicate more severe OCD symptoms.
Time Frame: Baseline (week 0), mid-treatment (week 6), end-of-treatment (week 12)
Population: Intent-to-treat analysis, which included all participants randomized to each treatment arm. Some participants dropped out prior to completion of the mid-treatment (week 6) or end-of-treatment (week 12) assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perspectives OCD | The Health and Well-Being Program
Number analyzed (Participants) | 60 | 60
score on a scale
  Week 0 | 25.12 (4.22) | 23.77 (4.60)
  Week 6: number analyzed (Participants) | 57 | 47
  Week 6 | 18.68 (5.34) | 20.49 (5.32)
  Week 12: number analyzed (Participants) | 57 | 46
  Week 12 | 16.14 (6.48) | 18.15 (5.67)
Statistical Analysis 1: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in Y-BOCS total scores between the treatment groups at endpoint (week 12); Test type: Superiority; p = 0.0871, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons because this was the pre-specified primary endpoint comparison. The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Mean Difference (Final Values) = -2.0475, 95% CI 2-sided [-4.3977 to 0.3027] — The effect is presented as the Perspectives OCD group outcome compared to the Health and Well-Being Program group outcome at the trial end-point (week 12)
Statistical Analysis 2: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in the change from baseline to end-of-treatment Y-BOCS total scores between the treatment groups; Test type: Superiority; p = 0.0036, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Difference in the amount of change = -3.4385, 95% CI 2-sided [-5.7394 to -1.1376] — The effect is presented as the difference in the amount of symptom reduction (week 12 - week 0) between Perspectives OCD and the Health and Well-Being Program group (i.e., a group difference in the amount of change over time)

2. Secondary Outcome: Difference in Depression at the End of Week 12
Description: The Quick Inventory of Depressive Symptomatology (Self-report; QIDS-SR) is a self-report measure of depressive symptoms consisting of 16 scale items with responses ranging from 0 to 3, including one suicide item (item #12). Total scores range from 0 to 27 with higher scores indicating greater depression severity. The measure is a well-validated, sensitive measure of symptom severity in depression.
Time Frame: Baseline (week 0), mid-treatment (week 6), end-of-treatment (week 12)
Population: This was an intent-to-treat analysis, which included all participants randomized to each treatment arm. Some participants dropped out prior to completion of the mid-treatment (week 6) or end-of-treatment (week 12) assessments (see participant flow chart); a few more did not complete self-rated questionnaires after completing clinician-rated assessments (Perspectives OCD: n=1 at week 6, n=4 at week 12; Health and Well-Being Program: n=2 at week 6, n=2 at week 12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perspectives OCD | The Health and Well-Being Program
Number analyzed (Participants) | 60 | 60
score on a scale
  Week 0 | 8.70 (4.53) | 8.27 (4.11)
  Week 6: number analyzed (Participants) | 56 | 45
  Week 6 | 7.23 (5.10) | 7.00 (4.20)
  Week 12: number analyzed (Participants) | 53 | 44
  Week 12 | 6.36 (4.60) | 6.84 (4.89)
Statistical Analysis 1: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in depression severity (QIDS-SR total scores) between the treatment groups at endpoint (week 12); Test type: Superiority; p = 0.3616, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Mean Difference (Final Values) = -0.8743, 95% CI 2-sided [-2.7666 to 1.0181] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in the change from baseline to end-of-treatment depression severity (QIDS-SR total scores) between the treatment groups; Test type: Superiority; p = 0.1973, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Difference in the amount of change = -1.3076, 95% CI 2-sided [-3.3014 to 0.6862] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Difference in Functional Impairment at the End of Week 12
Description: Functional impairment was assessed using the Work and Social Adjustment Scale (WSAS). This scale uses a Likert scale from 0 (not at all) to 10 (extremely) to assess impairment in a person's ability to function in terms of work, home management, leisure activities. Total scores total range from 0-40, where higher scores indicate greater impairment.
Time Frame: Week 0, Week 6, and Week 12
Population: This was an intent-to-treat analysis, which included all participants randomized to each treatment arm. Some participants dropped out prior to completion of the mid-treatment (week 6) or end-of-treatment (week 12) assessments (see participant flow chart); a few more did not complete self-rated questionnaires after completing clinician-rated assessments (Perspectives OCD: n=1 at week 6, n=4 at week 12; Health and Well-Being Program: n=1 at baseline, n=2 at week 6, n=1 at week 12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perspectives OCD | The Health and Well-Being Program
Number analyzed (Participants) | 60 | 60
score on a scale
  Week 0: number analyzed (Participants) | 60 | 59
  Week 0 | 20.57 (8.91) | 18.80 (7.70)
  Week 6: number analyzed (Participants) | 56 | 45
  Week 6 | 16.04 (9.07) | 16.43 (10.84)
  Week 12: number analyzed (Participants) | 53 | 45
  Week 12 | 12.38 (8.99) | 14.98 (9.97)
Statistical Analysis 1: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in functional impairment (WSAS total scores) between the treatment groups at endpoint (week 12); Test type: Superiority; p = 0.1289, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Mean Difference (Final Values) = -2.7992, 95% CI 2-sided [-6.4246 to 0.8262] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in the change from baseline to end-of-treatment functional impairment (WSAS total scores) between the treatment groups; Test type: Superiority; p = 0.0137, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Difference in the amount of change = -4.5704, 95% CI 2-sided [-8.1939 to -0.9468] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Difference in Quality of Life at the End of Week 12
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) is a self-report measure of subjective quality of life, containing Likert items ranging from 1 (Very Poor) to 5 (Very Good). Total scores are presented as a percentage of the maximum value (i.e., ranging from 0 to 100), with higher scores indicating greater quality of life).
Time Frame: Week 0, Week 6, and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of the scale maximum score
Arm/Group | Perspectives OCD | The Health and Well-Being Program
Number analyzed (Participants) | 60 | 60
percentage of the scale maximum score
  Week 0: number analyzed (Participants) | 60 | 59
  Week 0 | 56.63 (15.12) | 59.02 (14.79)
  Week 6: number analyzed (Participants) | 56 | 45
  Week 6 | 62.93 (15.79) | 62.54 (16.26)
  Week 12: number analyzed (Participants) | 53 | 45
  Week 12 | 66.87 (16.82) | 63.04 (16.26)
Statistical Analysis 1: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in quality of life (Q-LES-Q-SF percentage scores) between the treatment groups at endpoint (week 12); Test type: Superiority; p = 0.1796, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Mean Difference (Final Values) = 4.3953, 95% CI 2-sided [-2.0543 to 10.8448] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Perspectives OCD vs The Health and Well-Being Program; Null hypothesis: there is no significant difference in the change from baseline to end-of-treatment quality of life (Q-LES-Q-SF percentage scores) between the treatment groups; Test type: Superiority; p = 0.0400, Mixed Models Analysis — The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a first-order heterogeneous auto-regressive (ARH(1)) covariance structure; Difference in the amount of change = 6.7962, 95% CI 2-sided [0.3140 to 13.2785] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected every 6 weeks after the baseline visit, during the mid-treatment assessment visit (week 6) and the post-treatment visit (week 12). At these assessments, participants were probed for adverse events that occurred since the last adverse event assessment (usually 6 weeks prior).
Description: Participants were asked 4 questions about: (1) any major physical health problems or major physical injuries; (2) seeing a physical health or mental health provider for any reason; (3) any hospitalizations; or (4) any other major problems or concerns, all pertaining to the time since they were assessed last. Any "yes" resulted in further inquiries into specific adverse events.
Arm/Group | Perspectives OCD | The Health and Well-Being Program
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60
Other Adverse Events (participants affected / at risk) | 23/60 | 27/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perspectives OCD (N=60) | The Health and Well-Being Program (N=60)
Worsening of mental health resulting in inpatient hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perspectives OCD (N=60) | The Health and Well-Being Program (N=60)
Gastrointestinal problems including diarrhea, norovirus, Crohn's disease, acid reflux (Gastrointestinal disorders) | 4 (5) | 1 (1)
COVID-19 and/or flu (Infections and infestations) | 2 (2) | 6 (6)
arthritis, leg/foot pain, muscle spasms, muscle tension, herniated disc, tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
increased depression, anxiety, and/or irritability (Psychiatric disorders) | 5 (5) | 6 (7)
worsening of OCD symptoms (Psychiatric disorders) | 2 (2) | 4 (4)
stress and anxiety due to job, relationships, death of a loved one, or household problems (Social circumstances) | 10 (11) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT04136626/Prot_SAP_000.pdf